CLINICAL TRIAL: NCT00004144
Title: Phase I Study of Bryostatin 1 and Gemcitabine (Gemzar)
Brief Title: Bryostatin 1 Plus Gemcitabine in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067375; P30CA022453 (NIH); WSU-Z-2021; NCI-T99-0014
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — bryostatin 1; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bryostatin 1 & gemcitabine hydrochloride (Experimental)
  Interventions: Drug: bryostatin 1; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bryostatin 1
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of bryostatin 1 plus gemcitabine in treating patients who have advanced cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gemcitabine when given concurrently with bryostatin 1 to patients with advanced refractory cancer.
* Access the pattern of toxicity of this drug regimen in this patient population.
* Determine the objective response rate, duration of response, and overall survival in patients treated with this drug regimen.
* Determine the influence of bryostatin 1 on the pharmacokinetics of gemcitabine.

OUTLINE: This is a dose escalation study.

Patients receive gemcitabine IV over 30 minutes, immediately followed by bryostatin 1 IV over 24 hours, weekly for 3 weeks (days 1, 8, and 15). Treatment repeats every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of gemcitabine and bryostatin 1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxic effects.

PROJECTED ACCRUAL: Approximately 2-3 patients per month will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced cancer (except hematological cancers) for which there is no standard therapy or have failed standard therapies
* Measurable or evaluable disease
* Clinically controlled brain metastases allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 8.0 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (elevated bilirubin due to Gilbert's syndrome allowed if direct bilirubin normal)
* AST less than 2.5 times ULN

Renal:

* Creatinine normal

Cardiovascular:

* No active cardiac disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent bacterial infection requiring antibiotics
* No serious concurrent medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* At least 3 weeks since systemic cytotoxic chemotherapy (including gemcitabine) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapy allowed
* No concurrent hormonal therapy (excluding contraceptives, appetite stimulants, or replacement steroids)

Radiotherapy:

* At least 3 weeks since radiotherapy to large areas of active bone marrow and recovered
* No concurrent radiotherapy

Surgery:

* Recovered from prior major surgery

Other:

* No concurrent antiviral nucleosides
* At least 1 month since prior investigational agents
* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] El-Rayes BF, Gadgeel S, Shields AF, Manza S, Lorusso P, Philip PA. Phase I study of bryostatin 1 and gemcitabine. Clin Cancer Res. 2006 Dec 1;12(23):7059-62. doi: 10.1158/1078-0432.CCR-06-1419. PMID 17145828